CLINICAL TRIAL: NCT01964274
Title: Relevance of the Peripheral Cholinesterase-activity on Neurocognitive Dysfunctions in Surgical Patients
Acronym: CESARO
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Department of Anesthesiology and Intensive Care Medicine CVK/CCM, Charite - Universitätsmedizin Berlin, Germany, Charite University, Berlin, Germany
Other Study IDs: CESARO
Record Dates: First submitted 2013-10-15; First posted 2013-10-17 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Postoperative Delirium
Keywords: Nursing Delirium Screening Scale,; Acetylcholinesterase Activity
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Surgical patients: Adult male and female patients undergoing surgery

SUMMARY:
In this prospective, multicenter observational study the investigators capture the perioperative course of peripheral cholinesterase activity. The focus is the perioperative inflammation causing postoperative delirium. Therefore we measure the activity of Acetylcholine-Esterase and Butyrylcholine-Esterase in whole blood of adults in the perioperative context. Early postoperative delirium will be detected by Nu-DESC in the Recovery Room or the Postanaesthesia-Care-Unit. The course of the peripheral cholinesterase activity will be compared with the incidence of postoperative delirium and other clinical dysfunctions.

We follow up the patients for up to five years regarding Delirum, comorbidities and mortality data.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with age 18 years and above scheduled for surgery with planned stay in Recovery Room or Postanesthesia-Care-Unit
* Offered patient information and written informed consent
* In-hospital stay for at least 24 hours

Exclusion Criteria:

* Patients with known pseudocholinesterase deficiency
* Participation in prospective intervention studies during the study period
* Analphabetism
* Unability of German and English language use
* Anacusis or Hypoacusis with hearing aid device, Amaurosis
* Lacking willingness to save and hand out data within the study
* Accommodation in an institution due to an official or judicial order
* Coworker of the clinic (study center)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult, elective surgery patients of both gender
Sampling Method: Probability Sample
Enrollment: 815 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Postoperative Delirium | Participants will be followed in the sample period, an exspected average of three days
  Postoperative Delirium (measured by Nursing Delirium Screening Scale)

SECONDARY OUTCOMES:
Organ Dysfunctions | Participants will be followed in the sample period, an exspected average of three days
Concomitant medication | Participants will be followed in the three postoperative days sample period
  Concomitant medications from Anticholinergic Drug Scale (ADS)
Postoperative Pain | Participants will be followed in the three postoperative days sample period
  According to Numeric Rating Scale
Duration of Intensive Care Unit Stay | Participants will be followed in the sample period, an exspected average of seven days
Duration of Hospital Stay | Participants will be followed in the sample period, an exspected average of four weeks
Duration of Mechanical Ventilation | Participants will be followed in the sample period, an exspected average of 168 hours
Readmission rate | Participants will be followed in the sample period, an exspected average of four weeks
Hospital Treatment Data | Participations will be followed for the duration of the operation day, an exspected time average of eight hours
  Operation time, surgery, anaesthesia
Postoperative Mortality | Participants will be followed for the duration of the sample period an exspected average of five years
  Mortality (measured inhouse-mortality according to the patients´records and based on the data record according to §21 Krankenhausentgeltgesetz - (KHEntgG))
Postoperative Delirium | Participants will be followed in the sample period, an exspected average of five years
  Postoperative Delirium (measured by Diagnosis of Delirium according to the patients´records and based on the data record according to §21 Krankenhausentgeltgesetz -(KHEntgG))
Comorbidities | Participants will be followed in the sample period, an exspected average of five years
  Comorbidities based on the data record according to §21 Krankenhausentgeltgesetz - (KHEntgG)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Study Director — Department of Anesthesiology and Intensive Care Medicine, Campus Charité Mitte and Campus Virchow-Klinikum, Charité - Universitätsmedizin Berlin
Locations (9):
- Germany (9):
  - Department of Anesthesiology and Intensive Care Medicine, Campus Charité Mitte and Campus Virchow-Klinikum, Charité - Universitätsmedizin Berlin, Berlin
  - Department of Anesthesia, Klinik für MIC, Berlin
  - Clinic for Anaesthesiology, Intensive Care Medicine, Palliative Medicine and Pain Medicine, Berufsgenossenschaftliches Universitätsklinikum Bergmannsheil, Bochum
  - Department of Anesthesiology, Universitätsklinikum Heidelberg, Heidelberg
  - Department of Anesthesiology, Klinikum Großhadern of the Ludwig Maximilians University of Munich, München
  - Department of Anesthesiology, Universitätsklinikum Regensburg, Regensburg
  - Department of Anesthesiology, Universitätsklinikum Ulm, Ulm
  - Department of anesthesiology and intensive care medicine, Wetzlar
  - Department of Anaesthesia and Critical Care, Universitätsklinikum Würzburg, Würzburg

REFERENCES:
- [Result] Muller A, Olbert M, Heymann A, Zahn PK, Plaschke K, von Dossow V, Bitzinger D, Barth E, Meister M, Kranke P, Herrmann C, Wernecke KD, Spies CD. Relevance of peripheral cholinesterase activity on postoperative delirium in adult surgical patients (CESARO): A prospective observational cohort study. Eur J Anaesthesiol. 2019 Feb;36(2):114-122. doi: 10.1097/EJA.0000000000000888. PMID 30431498
- [Derived] Michels B, Holzamer A, Graf BM, Bredthauer A, Petermichl W, Muller A, Zausig YA, Bitzinger DI. Butyrylcholinesterase as a perioperative complication marker in patients after transcatheter aortic valve implantation: a prospective observational study. BMJ Open. 2021 Jul 6;11(7):e042857. doi: 10.1136/bmjopen-2020-042857. PMID 34230011